CLINICAL TRIAL: NCT00238992
Title: A Prospective, Randomized, Open Label, Multicenter Trial of EC-MPS With Steroid Withdrawal vs EC-MPS With Standard Steroid Regimen for the Prevention of Acute Rejection Episodes in de Novo Renal Transplant Recipients.
Brief Title: Study of Enteric-coated Mycophenolate Sodium (EC-MPS) With Steroid Withdrawal vs EC-MPS With Standard Steroid Regimen in de Novo Renal Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A2405ES01
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Kidney de Novo Transplant
Keywords: Kidney, de novo transplant, steroid withdrawal, adults, EC-MPS and cyclosporine

INTERVENTIONS:
Drug: Enteric-coated Mycophenolate sodium (EC-MPS)

SUMMARY:
All patients of the core study who are interested of being treated with EC-MPS will be included in an open-label extension study to collect further information on the long-term safety, tolerability and efficacy of this drug.

The purpose of this study is to evaluate the feasibility of steroid withdrawal in the setting of immunosuppression with a combination of EC-MPS, cyclosporine and steroids in de novo kidney allograft recipients.

ELIGIBILITY:
Inclusion Criteria

* Male or female patients undergoing first kidney transplant.
* Patients aged 18 -70 years.
* Patients receiving an ABO identical or compatible graft. Exclusion Criteria
* Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ other than kidney.
* Positive HBsAg test
* Pre-Transplant PRA >50% or historical PRA >75% Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 2002-12; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
biopsy proven acute rejection incidence at 1 year post-transplantation

SECONDARY OUTCOMES:
Incidence of biopsy proven acute rejection episodes at 6 months
Incidence of treated rejection episodes at 6 months and 1 year
Incidence of steroid-resistant episodes at 6 months and 1 year
Patient and graft survival at 1 year
Cardiovascular profile (as measured by Cholesterol, HbA1, Glucose, incidence of HTA)
Percentage of patients free from steroids at 6 months and 1 year
Treatment safety

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis